CLINICAL TRIAL: NCT05052112
Title: A Randomized, Placebo-controlled, Double-blind, Cross-Over Study to Evaluate the Efficacy of E-PR-01 on Activity Induced Joint Pain
Brief Title: Cross-Over Study to Evaluate the Efficacy of E-PR-01 on Activity Induced Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: EB/210504/VTZO/JP
Record Dates: First submitted 2021-09-09; First posted 2021-09-22 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-controlled, Double-blind, Cross-Over Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-PR-01 200mg (Active Comparator): Oral administration : One capsule to be taken after breakfast and one capsule before dinner for around 5 to 7 days
  Interventions: Other: E-PR-01; Other: E- PR-02
- E-PR-02 200mg (Placebo Comparator): Oral administration : One capsule to be taken after breakfast and one capsule before dinner for around 5 to7 days
  Interventions: Other: E-PR-01; Other: E- PR-02

INTERVENTIONS:
Other: E-PR-01 — Active arm
Other: E- PR-02 — Placebo arm

SUMMARY:
This Clinical trial study for the effect of a product E-PR-01 will be studied for its ability to attain rapid pain relief in the individuals suffering from exercise-induced knee joint pain, as well as determine its sustained effect on pain reduction over a treatment period of five days.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo controlled, cross-over study to explore the effect of a product E-PR-01 on joint pain. Approximately 50 participants aged between ≥ 20 and ≤ 60 years will be screened. At least 40 participants will be randomized, and the participants will be crossed over both the IP and placebo arms. A minimum of 32 participants must complete the study, after accounting for the screening failure and dropout /withdrawal rate of 20% each. The duration of each treatment for all the study participants will be 5 days, the washout period between each treatment period being 5 ± 2 days.

The total study period from the first start of treatment visit, inclusive of the washout and treatment periods, is estimated to be 15 days.

ELIGIBILITY:
Inclusion Criteria:

1. Physically active adults aged ≥20 and ≤60 years with history of knee joint pain aggravation on physical stress (walking, running, cycling etc.).
2. Body Mass Index (BMI) ≥ 20 and ≤ 29.9 kg/m2.
3. Participants with self-reported joint pain of ≥ 60 on 100 mm VAS scale after walking on treadmill using modified Naughton's protocol.
4. Participants with no or minimal pain at rest (≤ 30 mm on VAS scale).
5. Participants willing to complete all the study procedures including study-related questionnaires and tasks, and comply with the study requirements.
6. Participants willing to abstain from the restricted supplements and medications prior to inclusion and throughout the study period.
7. Participants with the ability to read and provide written, personally signed, and dated informed consent to participate in the study.

Exclusion Criteria:

1. Known cases of osteo-, rheumatic- or any other form of arthritis.
2. Participants fulfilling ≥ 3 of the following ACR criteria:

   i. Over the age of 50 years ii. Less than 30 minutes of morning stiffness iii. Crepitus on active motion iv. Bony tenderness v. Bony enlargement vi. No palpable warmth at the knee
3. Participants suffering from Insomnia and restless leg syndrome.
4. Participants with uncontrolled Hypertension, as characterized by Systolic Blood Pressure (SBP) >139 mmHg and Diastolic Blood Pressure >89 mmHg.
5. Participants currently on anti-hypertensives
6. Participants suffering from Type II Diabetes Mellitus.
7. Participants with history of lower limb injure in the past six months.
8. Participants currently on joint health supplements and medications.
9. Participants with a history of knee surgery, replacement, or any non-knee surgical procedures that may impact the study outcomes
10. Participants who have used Intraarticular injections in the last six months.
11. Participants who have undergone a significant cardiovascular event in the past six months.
12. Individuals with history of hyperacidity with at least one episode/ week.
13. Individuals with diagnosed cases of migraine.
14. History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic, or neurological disorders, that in the judgment of the investigator, would interfere with the participant's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the participant at undue risk.
15. Participants who have any other disease or condition, or are using any medication, that in the judgment of the investigator would put the participant at unacceptable risk for participation in the study or may interfere with evaluations in the study or noncompliance with treatment or visits.
16. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
17. Participants who have participated in a study of an investigational product 90 days prior to the screening.
18. Participants with heavy alcohol consumption, defined as For men: More than 14 standard alcoholic drink (SAD)/week or more than 4 SAD in a day.

    For women: More than 7 SAD/week or more than 3 SAD in a day.
19. Binge drinkers, defined as 4 or more SAD for women, and 5 or more SAD for men, in a 2-hour time frame.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Time to Meaningful pain relief assed by Visual Analogue scale | From baseline Day 1 for both treatment period
  To determine the effect of IP after single dose on time taken to achieve meaningful pain relief as assessed by the time taken to have a reduction of at least 40 % from baseline (0-hour post exertion) on a 100-point pain visual analogue scale as compared to placebo..

SECONDARY OUTCOMES:
Pain Intensity Difference (PID) | At Post IP 2 hour, 3 hour and 4 hours Day 1 of treatment 1 and Post IP 2 hour, 3 hour and 4 hours Day 1 of treatment 2
  In this study, the Pain VAS will be used as the method of pain intensity assessment. The values of Pain VAS measured right after IP consumption and each specified time intervals will be the value used to assess PID.at 2-, 3- and 4-hours Day 1 as compared to placebo. Minimum score is 0 represent No pain and 100 means worst possible pain.
Sum of Pain Intensity Difference SPID | at 0-hour post exertion and at 4 hours post IP Day 1 of treatment 1 and 0-hour post exertion and at 4 hours post IP Day 1 of treatment 2
  VAS score will be taken at 0-hour post exertion and at 4 hours post IP consumption after the performance of the modified Naughton Protocol. The summation of the PID values obtained will be used to calculate the sum of Pain Intensity Difference (SPID). Minimum score is 0 represent No pain and 100 means worst possible pain.
  SPID (ti-ti+n) = ∑ (PIDi)*(ti+1-ti)

CONTACTS AND LOCATIONS:
Locations (1):
- Vedic Lifesciences, Mumbai, Maharashtra, India